CLINICAL TRIAL: NCT02785211
Title: A Modified Behavioral Activation Treatment for Geriatric Depressive Symptoms in Left-behind Elderly in Rural China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S181
Record Dates: First submitted 2016-04-01; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Health Behavior; Depression
MeSH Terms: conditions — Health Behavior; Depression

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Behavioral Activation Treatment (Experimental): The modified model will be provided weekly to four groups for intervention, each group including about 10 participants with 1 facilitator for a period of 8 weeks after the baseline survey and general introduction. Each of the 8-week sessions will last for 2 hours. Groups 1 to 4 will have sessions on Mondays, Tuesdays, Wednesdays, and Thursdays respectively; four groups will meet on the same day of the week for all 8 weeks. The scheduling and timing of intervention provide consistency of scheduling for participants.
  Interventions: Behavioral: Behavioral Activation Treatment
- control group (Placebo Comparator): For the control group, participants will receive regular physical examinations and education by village doctors weekly during the 8 week intervention.The weekly visits for every old people whose age above 65 by country doctors are not arranged by our study, it is the country doctors" routine work by government health policy. This study was permitted by the local community health center, the director with specific responsibility will inform all country doctors to support our study.
  Interventions: Behavioral: Behavioral Activation Treatment

INTERVENTIONS:
Behavioral: Behavioral Activation Treatment — The modified model will be provided weekly to four groups for intervention, each group including about 10 participants with 1 facilitator for a period of 8 weeks after the baseline survey and general introduction. Each of the 8-week sessions will last for 2 hours. Groups 1 to 4 will have sessions on Mondays, Tuesdays, Wednesdays, and Thursdays respectively; four groups will meet on the same day of the week for all 8 weeks. The scheduling and timing of intervention provide consistency of scheduling for participants.

SUMMARY:
Background: It is essential to understand how to prevent and treat the epidemic of depression. Several studies have reported the prevalence of depressive symptoms in the urban population in China, but there is a lack of information regarding intervention for depression in rural left behind old elderly people.

Objective: To evaluate the effectiveness of a Modified Behavioral Activation Treatment (MBAT) Intervention on reducing depressive symptoms in rural left behind elderly people.

Methods: 80 rural left behind elderly people who had a Geriatric Depression Scale(GDS) score between 11 and 25 will be recruited and randomly assigned to the intervention (n=40) and control group(n=40). The intervention group will be received both MBAT and treatment-as-usual for 8 weeks while the control group received treatment-as-usual. Both groups will be assessed with the GDS, Beck Anxiety Inventory (BAI), and Oxford Happiness Questionnaire (OHQ) at baseline, immediately post-intervention, and at 3 months post-intervention.

Significance: This is the first time BA psychotherapy will be used in China.The current study will develop an intention model based on the traditional BA and CBT. The recurrence and seriousness of depression symptoms may be reduced by the intervention program. We hope that MBAT in clients will provide a direction for the management of mental health in rural left-behind elders..

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years of age;
* Only one participant from each family;
* Left-behind for longer than 6 months;
* GDS score between 11 and 25.

Exclusion Criteria:

* Psychiatric and medical comorbidities that are potentially life threatening or expected to severely limit client participation or adherence;
* Those who are currently seeing a cognitive behavioral therapist, psychotherapist or counselor;
* People unable to understand and fill out the questionnaires.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
depression assessed with the Geriatric Depression Scale | After 8 weeks MBAT, the GDS scores in the intervention group decreased significantly compared to those in the control group
  Depression symptoms will be measured using the validated Chinese version of the Geriatric Depression Scale. The scale consists of 30 questions, used to screen for depressive symptoms in community-dwelling elderly to evaluate the effect of reminiscence on depressive symptoms.Questions ask elderly participants to describe feelings over the past week and responses are "Yes" or "No". Its ease of use makes it suitable for community studies. Scores from 0 to 10 are regarded as normal, 11-20 as mild depression, 21-25 as moderate depression, and 26-30 as severe depression. The internal consistency reliability of the scale was 0.89 and test-retest reliability was 0.85; criterion related validity was 0.95, and parallel validity using the center for Epidemiologic Studies Depression Scale (CES-D) was 0.96 in Chinese participants (Wang,1999).

REFERENCES:
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Dimidjian S, Barrera M Jr, Martell C, Munoz RF, Lewinsohn PM. The origins and current status of behavioral activation treatments for depression. Annu Rev Clin Psychol. 2011;7:1-38. doi: 10.1146/annurev-clinpsy-032210-104535. PMID 21275642
- [Background] Dobson KS, Hollon SD, Dimidjian S, Schmaling KB, Kohlenberg RJ, Gallop RJ, Rizvi SL, Gollan JK, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the prevention of relapse and recurrence in major depression. J Consult Clin Psychol. 2008 Jun;76(3):468-77. doi: 10.1037/0022-006X.76.3.468. PMID 18540740